CLINICAL TRIAL: NCT03546140
Title: Diagnostic of Human Immunodeficiency Virus (HIV) and Other Sexual Transmission Diseases (STD) in High Risk Populations: Men Who Have Sex With Men (MSM) Users of Chemsex
Acronym: Care_ChemS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project manager Clinical Trials Unit, Fundacion Clinic per a la Recerca Biomédica
Other Study IDs: Care_ChemS_ClinC -001-2017
Record Dates: First submitted 2018-05-09; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and fixed tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to offer diagnostic tests for HIV, HCV and other STD in the risk group of men having sex with men (MSM) users of Chemsex

DETAILED DESCRIPTION:
The main objective is to offer diagnostic tests for HIV, HCV and other STD in the risk group (MSM users of Chemsex) with the purpose of conduct diagnosis, early treatment and monitoring of this infections and reduce the incidence rate of the same ones

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Men MSM/transgender referred from PEP office
* Men MSM/transgender referred from urgency service attended for acute intoxication or an STD
* Men MSM/transgender referred from STD office
* Men MSM/transgender referred from a local ONG attended for chemsex use
* Specifically drug use for having sexual relations, at least once in a month in the lasts 6 months or more than 10 times the last year
* Reading and understanding ability
* Patients should be given written informed consent
* Negative HIV and HCV men
* HIV positive men but HIC negative referred from HIV daily hospital
* Disposal of sanitary card from CatSalut

Exclusion Criteria:

* Men that not accomplish inclusion criteria
* Drug use for another purposes not sexual
* Drug use for having occasional sexual relations, least than once in the past 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men MSM that come from HIV, urgency service and other from the hospital and from a local ONG
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Number of HIV, | 2 years
  HIV positive serology
number of HCV seroconversion | 2 years
  HCV positive serology
number STD seroconversion | 2 years
  positive serology

SECONDARY OUTCOMES:
type of consumer drug | 2 years
  number and name ( Visual Analog Score for drug)
clinical outcomes | 2 years
  number of hospital admissions for acute intoxications
analytical outcomes | 2 years
  VDRL serology
analytical outcomes | 2 years
  PCR CT/GN(pharynx / urethra / anus)
weight | 2 years
  in kilograms